CLINICAL TRIAL: NCT04088175
Title: A Randomized, Open-Label, Cross-Over Study to Characterize Puffing Topography With Use of JUUL Electronic Nicotine Delivery Systems (ENDS) in Adult, Closed-System ENDS Consumers
Brief Title: Study to Characterize Puffing Topography With Use of JUUL Electronic Nicotine Delivery Systems (ENDS) in Adult, Closed-System ENDS Consumers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Collaborators: Los Angeles Clinical Trials (Unknown); Battelle Memorial Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PROT-00032
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2020-02

CONDITIONS: Electronic Cigarette Use
Keywords: Topography
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: Randomized, open label, 2-group, 4-period cross-over study in adult closed system ENDS consumers designed to evaluate puff topography parameters with use of JUUL ENDS products .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Virginia Tobacco and Menthol (Experimental): Subjects randomized to Group 1 will use JUUL ENDS Virginia Tobacco and Menthol flavors
  Interventions: Other: JUUL ENDS - Virginia Tobacco 5% nicotine strength; Other: JUUL ENDS - Virginia Tobacco 3% nicotine strength; Other: JUUL ENDS - Menthol 5% nicotine strength; Other: JUUL ENDS - Menthol 3% nicotine strength
- Group 2 - Mint and Mango (Experimental): Subjects randomized to Group 2 will use JUUL ENDS Mint and Mango flavors
  Interventions: Other: JUUL ENDS - Mint 5% nicotine strength; Other: JUUL ENDS - Mint 3% nicotine strength; Other: JUUL ENDS - Mango 5% nicotine strength; Other: JUUL ENDS - Mango 3% nicotine strength

INTERVENTIONS:
Other: JUUL ENDS - Virginia Tobacco 5% nicotine strength — JUUL ENDS - Virginia Tobacco 5% nicotine strength
  Arms: Group 1 - Virginia Tobacco and Menthol
Other: JUUL ENDS - Virginia Tobacco 3% nicotine strength — JUUL ENDS - Virginia Tobacco 3% nicotine strength
  Arms: Group 1 - Virginia Tobacco and Menthol
Other: JUUL ENDS - Menthol 5% nicotine strength — JUUL ENDS - Menthol 5% nicotine strength
  Arms: Group 1 - Virginia Tobacco and Menthol
Other: JUUL ENDS - Menthol 3% nicotine strength — JUUL ENDS - Menthol 3% nicotine strength
  Arms: Group 1 - Virginia Tobacco and Menthol
Other: JUUL ENDS - Mint 5% nicotine strength — JUUL ENDS - Mint 5% nicotine strength
  Arms: Group 2 - Mint and Mango
Other: JUUL ENDS - Mint 3% nicotine strength — JUUL ENDS - Mint 3% nicotine strength
  Arms: Group 2 - Mint and Mango
Other: JUUL ENDS - Mango 5% nicotine strength — JUUL ENDS - Mango 5% nicotine strength
  Arms: Group 2 - Mint and Mango
Other: JUUL ENDS - Mango 3% nicotine strength — JUUL ENDS - Mango 3% nicotine strength
  Arms: Group 2 - Mint and Mango

SUMMARY:
A randomized, open label, 2-group, 4-period cross-over study in adult closed system ENDS consumers designed to evaluate puff topography parameters with use of JUUL ENDS products (Virginia Tobacco, Menthol, Mint, and Mango flavors, each at 5% and 3% nicotine strengths).

DETAILED DESCRIPTION:
Subjects who successfully complete screening procedures, including a brief trial with each of the JUUL flavors at the 5% strength, will be eligible to participate in the study.

Subjects will be randomized into one of two (2) groups (Virginia Tobacco and Menthol or Mint and Mango, each at both nicotine strengths) and to one of four (4) product use sequences specifying the order for which they will use the assigned products.

Apart from the final in-clinic visit, study visits will include two puff topography sessions; each session will be separated by 2 hours (minimum) after completion of the previous topography session. Puff topography sessions will include 1 hour of ad libitum product use according to the subject's usual ENDS product use procedures. A Baseline topography session will be done using the subject's usual ENDS product to provide context to the JUUL results. The Baseline session will be followed by a topography session with a JUUL product. Subsequent clinic visits will include two different JUUL products: (1) The JUUL product used during the current study period and (2) The JUUL product for the next study period. The final in-clinic visit will only include one puff topography session with the JUUL product used during the final study period.

Puff topography measurements will be collected with a Clinical Research Support System (CReSS) device. Subjects who present with a preferred ENDS product that is not compatible with adapters fitting the CReSS device will participate in the 1 hour product use session without using the CReSS device. The weight of the product (pod/cartomizer without the battery; resolution of 0.1 mg) will be measured before and after use.

Subjects will complete subjective effects questionnaires (Product Liking and PES) after completion of each topography session. The subjective effects questionnaires and product use data will be used to assess potential factors that might impact the puff topography parameters.

After completion of required study events at each clinic visit, subjects will be discharged with a 7-day supply of the appropriate JUUL product and with instructions that the provided product is the only tobacco/nicotine containing product that they are to use, and to reach out to the clinic if it appears that they will run out of JUUL products before the next clinic visit. Subjects will be also be asked to complete an at-home product use log each day until returning to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Provides voluntary consent to participate in this study documented on the signed informed consent form (ICF).
2. Male or female, 21 to 65 years of age, inclusive, at Screening.
3. Has been a closed system ENDS consumer for at least 3 months prior to Screening.
4. Currently consumes at least half a pod or cartomizer e-liquid per day as reported at Screening.
5. Has a positive urine cotinine (≥200 ng/mL) at Screening.
6. Has an exhaled CO <8 ppm at Screening.
7. A female subject of childbearing potential must have been using 1 of the following forms of contraception, and agree to continue using it through completion of the study:

   hormonal (e.g., oral, vaginal ring, transdermal patch, implant, or injection) consistently for at least 3 months prior to Screening; double barrier method (e.g., condom with spermicide, diaphragm with spermicide) at Screening; intrauterine device for at least 3 months prior to Screening; a partner who has been vasectomized for at least 6 months prior to Screening; abstinence beginning at least 6 months prior to Screening.
8. A female subject of non childbearing potential must be postmenopausal with amenorrhea for at least 1 year prior to Screening and follicle stimulating hormone (FSH) levels consistent with postmenopausal status or have undergone one of the following sterilization procedures at least 6 months prior to Screening:

   hysteroscopic sterilization; bilateral tubal ligation or bilateral salpingectomy; hysterectomy; bilateral oophorectomy.
9. Is willing to comply with the requirements of the study, including a willingness to use the study products during the study.

Exclusion Criteria:

1. Has a history or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Has a clinically significant abnormal finding on the physical examination, medical history, vital signs, ECG, or clinical laboratory results, in the opinion of an Investigator.
3. Has had an acute illness (e.g., upper respiratory infection, viral infection) requiring treatment within 14 days prior to Baseline.
4. Has a fever (>100.5°F) at Screening or Baseline.
5. Has a body mass index (BMI) >40.0 kg/m2 or <18.0 kg/m2 at Screening.
6. Has a history of drug or alcohol abuse within 24 months of Screening, as determined by the Investigator.
7. Has or has a history of diabetes mellitus, asthma, or chronic obstructive pulmonary disease.
8. Has a systolic blood pressure <90 or >150 mmHg, diastolic blood pressure <40 or >95 mmHg, or heart rate <40 or >99 bpm at Screening.
9. Has experienced an allergic reaction following previous e-cigarette use or with exposure to any primary components of the e-liquids (nicotine, flavor, benzoic acid, propylene glycol and glycerol).
10. Has a positive urine screen for alcohol or drugs of abuse at Screening or Baseline.
11. If female, the subject is pregnant, has a positive urine pregnancy test at screening, is lactating, or intends to become pregnant during the time period from screening through the end of study.
12. Has used any nicotine-containing product other than closed-system ENDS products (e.g., cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) within 14 days prior to Baseline.
13. Has used any prescription cessation treatments, including, but not limited to, varenicline (Chantix®) or bupropion (Zyban®) within 3 months prior to Screening.
14. Negative response (i.e., unwilling to use or unable to tolerate; e.g., experiences AEs during the product trial that will prevent the subjects from continuing to use the study products as judged by the Investigator) to any of the JUUL products at Screening.
15. Is a self-reported puffer (i.e., draws aerosol into the mouth and throat but do not inhale).
16. Is planning to quit ENDS product use during the study or postponing (within 30 days of screening) a quit attempt in order to participate in the study.
17. Has participated in a previous clinical study for an investigational drug, device, biologic, or tobacco product within 30 days prior to Screening.
18. Is or has a first-degree relative (i.e., parent, sibling, child) who is a current employee of the study site.
19. Is or has a first-degree relative (i.e., parent, sibling, child) who is a current employee, shareholder, or is member of the board of directors of JUUL Labs Inc.
20. Has previously taken part in, has been excluded or withdrawn from, or has completed this study.
21. In the opinion of the Investigator, the subject should not participate in this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Puff Topography Parameter - Puff Duration | 29 Days
  To characterize post-acclimatization mean and total puff duration
Puff Topography Parameter - Puff Volume | 29 Days
  To characterize post-acclimatization mean and total puff volume
Puff Topography Parameter - Flow Rate | 29 Days
  To characterize post-acclimatization mean and peak puff flow rate
Puff Topography Parameter - Inter-puff interval | 29 Days
  To characterize post-acclimatization mean and total inter-puff interval
Puff Topography Parameter - Number of Puffs | 29 Days
  To characterize post-acclimatization total number of puffs

SECONDARY OUTCOMES:
Product Use - Product Weight Changes | 29 Days
  To measure product weight changes during each puff topography session
Product Use - Number of Pods Started Each Day | 29 Days
  To measure number of pods started each day during the ambulatory period
Product Use - Number of Puffs Per Day | 29 Days
  To measure number of puffs per day during the ambulatory period
Subjective Measure of product liking | 29 Days
  To assess the relationship between puff topography parameters and JUUL ENDS liking using a "Product Liking Questionnaire". Visual analogue scale with scale 0 (Not at all) to 100 (A Great Deal) in response to the instruction "Please indicate on the line below how much you liked the electronic cigarette product you used during this topography session."
Subjective Measure of product evaluation | 29 Days
  To assess the relationship between puff topography parameters and JUUL ENDS product evaluation using a "Modified Product Evaluation Scale". Scale consists of 21 questions that are categorized into four multi-item sub-scales: (1) "Satisfaction" (items 1, 2, 3, and 12); (2) "Psychological Reward" (items 4 through 8); (3) "Aversion" (items 9, 10, 16, and 18); and (4) "Relief" (item 11, 13, 14, 15, and reversed for item 20). Items 17 and 21 will be summarized individually.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Los Angeles Clinical Trials, Burbank, California
  - Battelle Public Health Lab, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD to other researchers.